CLINICAL TRIAL: NCT02237001
Title: A Prospective, Non-randomized, Multi-Center Investigation of All-suture-based Repair of Horizontal Meniscal Tears (STITCH Study)
Brief Title: Study of Suture Repair of Torn Meniscus in the Knee
Acronym: STITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTX-CP001
Record Dates: First submitted 2014-09-06; First posted 2014-09-11 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Meniscal Tear; Meniscus Tear
Keywords: meniscal; meniscus; repair; knee; arthroscopy knee; horizontal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Suture-based meniscal repair
  Interventions: Device: Suture-based meniscal repair

INTERVENTIONS:
Device: Suture-based meniscal repair — Suture-based meniscal repair

SUMMARY:
Horizontal meniscus tears meeting specified criteria will be repaired by any commonly used suture technique. Subjects will be followed for 2 years to evaluate the effectiveness of the repair, by assessing the re-operation rate, and by assessing improvements in knee pain and knee function.

DETAILED DESCRIPTION:
Potential subjects will undergo Screening for eligibility based on Inclusion/Exclusion criteria. Screening will include an x-ray of the injured knee and evaluation of an MRI of the injured knee within 6 months prior to the scheduled procedure. During the procedure, the meniscal tear will be evaluated by arthroscopy to determine if the tear meets study requirements. If the meniscal tear is determined to meet inclusion/exclusion criteria, the subject will be considered enrolled. If any inclusion/exclusion criteria is not met, the subject will be considered a screen failure and will not be enrolled. For enrolled subjects, specific information regarding the repair and repair technique will be collected during the procedure, including still and video images.

Subjects will be contacted 7-15 days post-procedure for safety follow-up. Subjects will return for follow-up visits at approximately post-procedure Days 90, 185, 365 and 730. Identical questionnaires will be completed at each visit to assess knee pain and knee function. Safety information will be collected at each post-procedure visit. Additionally, an in-office arthroscopy of the treated knee will be performed at participating sites at Day 185, an MRI of the treated knee will be performed at Day 365 and an X-ray of the treated knee will be performed at Day 730. The patient will exit the study at the Day 730 visit.

ELIGIBILITY:
Screening Inclusion Criteria:

Subjects of either gender may be eligible for inclusion in the study only if they meet all of the following criteria:

* Able and willing to give informed consent by voluntarily providing written informed consent in accordance with governing Institutional Review Board
* 18 to 60 years of age, inclusive at the time of screening;
* History indicative of meniscal pathology (e.g., pain, mechanical symptoms described as locking, clicking or giving way);
* Physical exam consistent with meniscus tear (e.g., locked joint, joint line tenderness and/or pain on meniscal compression);
* If prior ligament reconstruction, the study knee is clinically stable;
* Preoperative MRI evidence within 6 months consistent with a horizontal/radial/oblique meniscus tear in the symptomatic compartment

Arthroscopy Inclusion Criteria:

Consented subjects may be included in the study only if, upon arthroscopic inspection, their meniscal study lesion meets all of the following criteria established by the International Society of Arthroscopy, Knee Surgery and Orthopaedic Sports Medicine (ISAKOS) (see Appendix 1):

* Zone location: circumferential location of tear includes locations within 10mm of the peripheral rim of the meniscus;
* Radial location: any location from anterior to posterior;
* Tear pattern: primarily horizontal or oblique in orientation (not to exceed 45 degrees from horizontal);
* Compartment: either lateral or medial, but not both;
* Opposite compartment meniscal tear (if present) limited to the central portion (i.e., Zone 3/"white zone");
* Tear amenable to repair with all suture-based techniques.

Screening Exclusion Criteria:

Subjects will be excluded from the study for any of the following reasons:

* Arthritis in the study knee (Kellgren-Lawrence Grade 3 or higher [See Appendix 4]);
* Body Mass Index (BMI) ≥35 kg/m2;
* Previous meniscal repair or meniscectomy of the study meniscus;
* Unstable knee;
* Malalignment (> 5 degrees) of the study knee, based on X-ray within 6 months requiring osteotomy and/or requiring correction;
* History of constitutional/systemic inflammatory/arthritic problem or pain condition, history of knee infection, vascular condition of legs, benign neoplasms of knee, hepatitis, HIV, drug/alcohol abuse, tobacco use, cancer;
* Expected to undergo any other primary treatment of the knee;
* Any concomitant painful or disabling disease, condition or post-procedure status of either lower extremity that would interfere with evaluation or rehabilitation of the study knee.
* Pregnant or planning to become pregnant in the next 2 years.

Arthroscopy Exclusion Criteria:

Subjects will be excluded from the study if their study meniscus lesion meets any of the following criteria at arthroscopy:

* Tear pattern: primarily vertical longitudinal in orientation;
* Partial meniscectomy of any portion of the study meniscus extends beyond the central portion (i.e., Zone 3/"white zone");
* Intact or partially intact meniscus tear that, in the opinion of the Investigator, does not require repair;
* Poor meniscal tissue quality such that it will not hold a suture;
* Any portion of the meniscus repair that, in the opinion of the Investigator, is best treated using an implant other than suture;
* Bicompartmental Zone 1/"red zone" and/or Zone 2/"red-white zone" meniscal tears;
* Performance of a significant concomitant procedure intended as a therapeutic intervention on the study knee;
* Arthritis in the surgical knee (International Cartilage Research Society [ICRS] Grade 3b or higher or Modified Outerbridge Grade III or higher)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Kurzweil, MD, Principal Investigator — Memorial Orthopedic Surgical Group Long Beach; Darvin Griffin, Study Chair — Smith & Nephew, Inc.
Locations (8):
- United States (8):
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Memorial Orthopedic Surgical Group Long Beach, Long Beach, California
  - Andrews Research and Education Foundation, INC, Gulf Breeze, Florida
  - OrthoIndy South, Greenwood, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Winchester Medical Center, Winchester, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurzweil PR, Lynch NM, Coleman S, Kearney B. Repair of horizontal meniscus tears: a systematic review. Arthroscopy. 2014 Nov;30(11):1513-9. doi: 10.1016/j.arthro.2014.05.038. Epub 2014 Aug 6. PMID 25108905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled at clinics from 19NOV2014 until 08NOV2017; last subject visit was 18NOV2019
Pre-assignment Details: The planned sample size of 30 subjects was accrued for the Safety Population (SAF); however, a total of 4 subjects were excluded to comprise the Analysis Population (AS) due to late screen failure (eligibility criteria) or withdrawal by the subject.
Period: Overall Study
Arm/Group | Treatment
Started | 30
6 Month Follow-up | 27
12 Month Follow-up | 21
24 Month Follow-up | 19
Completed | 19
Not Completed | 11
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Eligibility criteria/Late Screen Failure | 3
Not completed — Re-operation | 4
Not completed — Incarceration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 24
  Ethnicity: Hispanic | 2
  Ethnicity: Asian | 2
  Ethnicity: Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 30
Height [Mean (Standard Deviation); unit: inches] | 69.25 (3.897)
Weight [Mean (Standard Deviation); unit: pounds (lb)] | 176.68 (33.356)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.68 (3.502)
Body Mass Index (BMI) Group [Count of Participants; unit: Participants]
  <30 | 26
  >=30 | 4

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Re-operation of the Index Meniscus Repair Site (Incidence of Subjects Requiring Re-operation)
Description: Occurrence of any re-operation of study knee to treat previously repaired meniscal tear during the 2 years following the study procedure.
Time Frame: 6 months, 1 year, and 2 years
Population: Overall number of participants analyzed indicates total number of participants enrolled in the Safety Population (SAF) at 6 months that provided data. Number analyzed for each time frame indicates all data available starting at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 27
Participants
  Freedom from re-operation at 6 months: Participants Free From Re-operation | 26
  Freedom from re-operation at 6 months: Participants Requiring Re-operation | 1
  Freedom from re-operation at 1 year: number analyzed (Participants) | 25
  Freedom from re-operation at 1 year: Participants Free From Re-operation | 23
  Freedom from re-operation at 1 year: Participants Requiring Re-operation | 2
  Freedom from re-operation at 2 years: number analyzed (Participants) | 23
  Freedom from re-operation at 2 years: Participants Free From Re-operation | 19
  Freedom from re-operation at 2 years: Participants Requiring Re-operation | 4

2. Secondary Outcome: Change in Knee Pain and Function by Completion of International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC Knee Evaluation) at 3 Months, 6 Months, 1 Year, and 2 Years
Description: Change in knee pain and function will be measured by completion of The International Knee Documentation Committee (IKDC) Subjective score. The IKDC Score was developed to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment, including patients with meniscal injuries.
  There are three domains: 1) symptoms, including pain, stiffness, swelling, locking/catching, and giving way (7 items), 2) sports and daily activities (10 items), and 3) current knee function and knee function prior to knee injury (1 item, not included in the score). Responses vary for each item. The possible score ranges from 0-100, where 100 = no limitation with daily or sporting activities and the absence of symptoms.
Time Frame: Baseline, 3 months, 6 months, 1 year, and 2 years
Population: 30 participants in Safety Population (SAF) and 26 participants in Analysis Population (AS). Planned sample size of 30 participants was accrued for SAF; however, a total of 4 participants were excluded to comprise AS due to late screen failure or withdrawal by participant. Each row represents all enrolled participants at the referenced time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  IKDC Baseline | 36.7 (16.2)
  IKDC Change from Baseline at 3 months: number analyzed (Participants) | 24
  IKDC Change from Baseline at 3 months | 23.9 (24.1)
  IKDC Change from Baseline at 6 months: number analyzed (Participants) | 24
  IKDC Change from Baseline at 6 months | 32.3 (25.1)
  IKDC Change from Baseline at 1 year: number analyzed (Participants) | 21
  IKDC Change from Baseline at 1 year | 40.8 (21.0)
  IKDC Change from Baseline at 2 years: number analyzed (Participants) | 19
  IKDC Change from Baseline at 2 years | 41.8 (21.0)

3. Secondary Outcome: Change in Knee Pain and Function by the Knee Injury and Osteoarthritis Outcome Score (KOOS): Pain Score at 3 Months, 6 Months, 1 Year, and 2 Years
Description: Change in knee pain and function will be measured by completion the Knee Injury and Osteoarthritis Outcome Score (KOOS). There are five patient-relevant subscales of the KOOS, and each are scored separately: Pain (9 items), ADL function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items).
  A Likert scale is used and all items have five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the 5 scores is calculated as the sum of the items included and then each score is transformed to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no knee problems as common in orthopedic assessment scales and generic measures. An aggregate score is not calculated so that each of the 5 dimensions can be assess separately.
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  Pain Score Baseline | 52.2 (19.1)
  Pain Score Change from Baseline at 3 months: number analyzed (Participants) | 24
  Pain Score Change from Baseline at 3 months | 26.9 (26.2)
  Pain Score Change from Baseline at 6 months: number analyzed (Participants) | 24
  Pain Score Change from Baseline at 6 months | 26.8 (23.0)
  Pain Score Change from Baseline at 1 year: number analyzed (Participants) | 21
  Pain Score Change from Baseline at 1 year | 32.9 (20.0)
  Pain Score Change from Baseline at 2 years: number analyzed (Participants) | 19
  Pain Score Change from Baseline at 2 years | 31.4 (22.1)

4. Secondary Outcome: Change in Daily Living (ADL) Score at 3 Months, 6 Months, 1 Year, and 2 Years
Description: as for outcome 3
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  ADL Score Baseline | 58.4 (21.7)
  ADL Score Change from Baseline at 3 months: number analyzed (Participants) | 24
  ADL Score Change from Baseline at 3 months | 25.4 (24.0)
  ADL Score Change from Baseline at 6 months: number analyzed (Participants) | 24
  ADL Score Change from Baseline at 6 months | 26.1 (20.0)
  ADL Score Change from Baseline at 1 year: number analyzed (Participants) | 21
  ADL Score Change from Baseline at 1 year | 31.7 (18.2)
  ADL Score Change from Baseline at 2 years: number analyzed (Participants) | 19
  ADL Score Change from Baseline at 2 years | 28.9 (20.1)

5. Secondary Outcome: Change in Knee Pain and Function by the Knee Injury and Osteoarthritis Outcome Score (KOOS): Sport and Recreation Function (Sport) Score at 3 Months, 6 Months, 1 Year, and 2 Years
Description: as for outcome 3
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  Sport Score Baseline | 29.6 (21.9)
  Sport Score Change from Baseline at 3 months: number analyzed (Participants) | 22
  Sport Score Change from Baseline at 3 months | 22.9 (34.1)
  Sport Score Change from Baseline at 6 months: number analyzed (Participants) | 24
  Sport Score Change from Baseline at 6 months | 33.0 (36.3)
  Sport Score Change from Baseline at 1 year: number analyzed (Participants) | 21
  Sport Score Change from Baseline at 1 year | 46.8 (31.3)
  Sport Score Change from Baseline at 2 years: number analyzed (Participants) | 19
  Sport Score Change from Baseline at 2 years | 48.7 (31.2)

6. Secondary Outcome: Change in Knee Pain and Function by the Knee Injury and Osteoarthritis Outcome Score (KOOS): Symptom Score at 3 Months, 6 Months, 1 Year, and 2 Years
Description: as for outcome 3
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  Symptom Score Baseline | 56.3 (19.5)
  Symptom Score Change from Baseline at 3 months: number analyzed (Participants) | 24
  Symptom Score Change from Baseline at 3 months | 19.6 (30.3)
  Symptom Score Change from Baseline at 6 months: number analyzed (Participants) | 24
  Symptom Score Change from Baseline at 6 months | 21.0 (23.7)
  Symptom Score Change from Baseline at 1 year: number analyzed (Participants) | 21
  Symptom Score Change from Baseline at 1 year | 28.4 (20.8)
  Symptom Score Change from Baseline at 2 years: number analyzed (Participants) | 19
  Symptom Score Change from Baseline at 2 years | 28.4 (23.9)

7. Secondary Outcome: Change in Knee Pain and Function by the Knee Injury and Osteoarthritis Outcome Score (KOOS): Quality of Life (QOL) Score at 3 Months, 6 Months, 1 Year, and 2 Years
Description: as for outcome 3
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  QOL Score Baseline | 28.1 (18)
  QOL Score Change from Baseline at 3 months: number analyzed (Participants) | 24
  QOL Score Change from Baseline at 3 months | 27.6 (29)
  QOL Score Change from Baseline at 6 months: number analyzed (Participants) | 24
  QOL Score Change from Baseline at 6 months | 32.8 (28.4)
  QOL Score Change from Baseline at 1 year: number analyzed (Participants) | 21
  QOL Score Change from Baseline at 1 year | 42.0 (26.5)
  QOL Score Change from Baseline at 2 years: number analyzed (Participants) | 19
  QOL Score Change from Baseline at 2 years | 43.8 (27.2)

8. Secondary Outcome: Change in Knee Pain and Function by Lysholm Knee Questionnaire at 3 Months, 6 Months, 1 Year, and 2 Years
Description: Change in knee pain and function will be measured by completion of the Lysholm Knee Questionnaire. This tool measures the domains of symptoms and complaints and functioning of daily activities. The scale consists of 8 item and is scaled from 0 to 100, with a higher score indicating fewer symptoms and higher level of functioning.
Time Frame: Baseline, 3 months, 6 months, 1 year, and 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  Lysholm Score Baseline | 50.2 (17.6)
  Lysholm Score Change from Baseline at 3 months: number analyzed (Participants) | 24
  Lysholm Score Change from Baseline at 3 months | 21.3 (27.8)
  Lysholm Score Change from Baseline at 6 months: number analyzed (Participants) | 24
  Lysholm Score Change from Baseline at 6 months | 25.4 (23.9)
  Lysholm Score Change from Baseline at 1 year: number analyzed (Participants) | 21
  Lysholm Score Change from Baseline at 1 year | 30.9 (24.3)
  Lysholm Score Change from Baseline at 2 years: number analyzed (Participants) | 19
  Lysholm Score Change from Baseline at 2 years | 32.5 (22.2)

9. Secondary Outcome: Change in Knee Pain and Function by Tegner Activity Scale at 3 Months, 6 Months, 1 Year, and 2 Years
Description: Change in knee pain and function will be measured by completion of the Tegner activity scale. The Tegner activity scale was designed as a score of activity level to complement other functional scores for patients with ligamentous injuries. The Tegner activity scale is a numerical scale ranging from 0 to 10. Each value indicates the ability to perform specific activities. An activity level of 10 corresponds to participation in competitive sports, including soccer, football, and rugby at the elite level; an activity level of 6 points corresponds to participation in recreational sports; and an activity level of 0 is assigned if a person is on sick leave or receiving a disability pension because of knee problems. An activity level of 5 to 10 is recorded only if the patient participates in recreational or competitive sports.
Time Frame: Baseline, 3 months, 6 months, 1 year, and 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 26
score on a scale
  Tegner Score Baseline | 3.3 (2.4)
  Tegner Score Change from Baseline at 3 months: number analyzed (Participants) | 24
  Tegner Score Change from Baseline at 3 months | 0.2 (2.1)
  Tegner Score Change from Baseline at 6 months: number analyzed (Participants) | 24
  Tegner Score Change from Baseline at 6 months | 1.3 (3.3)
  Tegner Score Change from Baseline at 1 year: number analyzed (Participants) | 21
  Tegner Score Change from Baseline at 1 year | 1.8 (2.6)
  Tegner Score Change from Baseline at 2 years: number analyzed (Participants) | 19
  Tegner Score Change from Baseline at 2 years | 1.7 (2.5)

ADVERSE EVENTS:
Time Frame: Enrollment through end of study (2 years)
Description: Adverse events were collected & reported as complications per the protocol. A complication was any untoward medical occurrence, unfavorable and unintended sign (including clinically significant abnormal laboratory finding), symptom, or condition experienced by the subject and temporally associated with the procedure whether or not considered related to the procedure. The Sponsor then reviewed all AEs and classified per ISO, using the higher level of classification, whether it be Site or Sponsor.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Further non-repairable tear meniscus (Musculoskeletal and connective tissue disorders) | 1 (1)
Swelling in knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee repair did not heal (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30)
Neuropathy (Nervous system disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Swelling of knee (Musculoskeletal and connective tissue disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
No limitations reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2014-12-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT02237001/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT02237001/SAP_001.pdf